CLINICAL TRIAL: NCT06795698
Title: The Effect of Prophylactic Anticoagulation on Major Bleeding Events in Hospitalized Chronic Kidney Disease and Lower Limb Fracture Patients. a Phase 2, Randomized, Doble Blind, Control Trial
Brief Title: The Effect of Prophylactic Anticoagulation on Major Bleeding Events in Hospitalized Chronic Kidney Disease and Lower Limb Fracture Patients.
Acronym: FAA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Jonathan Samuel Chavez Iñiguez, Head of nephrology, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 257/18
Record Dates: First submitted 2024-12-28; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Fractures, Bone; CKD Stage 4; CKD Stage 3; CKD Stage 5; Enoxaparin Adverse Reaction; Anticoagulant-induced Bleeding; Thromboses, Venous
Keywords: chronic kidney disease; anticoagulation; bleeding; bone fracture; thrombosis
MeSH Terms: conditions — Fractures, Bone; Renal Insufficiency, Chronic; Venous Thrombosis; Hemorrhage; Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: two groups recieved anticoagulation or placebo since randomization
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding was achieved by shielding the patients from seeing the preparation of the study drug and having unblinded study personnel not involved in any study outcome assessments responsible for preparing and administering the study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anticoagulation (Active Comparator): The intervention drug of interest was prophylactic anticoagulation with enoxaparin 1mg/kg of ideal body weight subcutaneous every 24 hours in patients with eGFR <30ml/min/1.73m2 (REF); enoxaparin will continue till surgery, any mandatory adverse event, dead or discharge. Enoxaparin or placebo started on admission to the trial, stopped 12 hours before surgery and all patients received prophylaxis anticoagulation restarted 6 to 12 hours postoperatively according to orthopedic surgeon practices. We choose enoxaparin, a low molecular weight heparin according to the ACCP guidelines as the gold standard for VTE prophylaxis in orthopedic patients
  Interventions: Drug: Enoxaparin
- No anticoagulation (Placebo Comparator): The no anticoagulation strategy was considerate the control group, we choose as placebo a bolus of 10ml normal saline 0.9%, was prepared and administered behind a screen or curtain, and the drug was administered through normal IV tubes
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — enoxaparin 1mg/kg of ideal body weight subcutaneous every 24 hours in patients with eGFR <30ml/min/1.73m2

SUMMARY:
the risk of bleeding may be greater than the benefit of antithrombotic protection when prophylactically anticoagulating a patient with a lower limb fracture and advanced CKD.

The primary objective was to evaluate the risk major bleeding in patients with lower limb fractures and advance CKD. The secondary objectives were to assess major bleeding in patients with lower limb fractures in CKD stage 4 and 5, thrombosis, death.

ELIGIBILITY:
Inclusion Criteria:

* lower limb fracture before surgery
* CKD (chonic kidney disease)

Exclusion Criteria:

* <18 years old
* kidney transplant
* hospital stay <48 hours
* had received any anticoagulant before random assignment to a patient group
* had missing data that would render analysis incomplete

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Major bleeding | From date of randomization until the date of first documented major bleeding or death from any cause, whichever came first up to 20 days. From date of randomization until surgery. Pre-intervention/procedure/surgery.
  Number of Participants with Major bleeding were defined according to the International Society on Thrombosis and Haemostasis (ISTH) criteria (Schulman S). Defined as the composed event of: 1- Fatal bleeding, and/or; 2- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or; 3- Bleeding causing a fall in hemoglobin level of 2.0 g/dL or more, or leading to transfusion of two or more units of whole blood or red cells

SECONDARY OUTCOMES:
Thrombosis | From date of randomization until the date of first documented thrombosis, or date of death from any cause, whichever came first, assessed from date of randomization until surgery up to 20 days. Pre-intervention/procedure/surgery.
  Number of Participants with Thrombosis was defined as the occurrence of a definite or probable venous thromboembolism (VTE) event. As deep vein thrombosis (DVT) typically presents with pain, swelling, warmth, or erythema of the affected limb
Dead | through study completion, an average of 3 weeks
  Number of Participants dead
number of transfusions | From date of randomization until the date of first documented transfusions and number of transfusions. Pre-intervention/procedure/surgery.
  Number of transfusions presurgery
acute kidney injury | From date of randomization until the date of first documented acute kidney injury up to 20 days. From date of randomization until surgery. Pre-intervention/procedure/surgery.
  Number of Participants with acute kidney injury, defined as an increses in serum creatinine >0.3mg/dL during 48 hours period
hospitalization days | number of days in hospital. through study completion, an average of 3 weeks
  number of days in hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Civil de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The files and data are in the physical and electronic archives of the Civil Hospital of Guadalajara Fray Antonio Alcalde and can be requested with prior authorization. All data generated or analyzed during this study are included in this article. Further inquiries can be directed to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: for 5 years
Access Criteria: The files and data are in the physical and electronic archives of the Civil Hospital of Guadalajara Fray Antonio Alcalde and can be requested with prior authorization. All data generated or analyzed during this study are included in this article. Further inquiries can be directed to the corresponding author.

REFERENCES:
- [Background] Lieberman JR, Bell JA. Venous Thromboembolic Prophylaxis After Total Hip and Knee Arthroplasty. J Bone Joint Surg Am. 2021 Aug 18;103(16):1556-1564. doi: 10.2106/JBJS.20.02250. PMID 34133395
- [Background] Naylor KL, McArthur E, Leslie WD, Fraser LA, Jamal SA, Cadarette SM, Pouget JG, Lok CE, Hodsman AB, Adachi JD, Garg AX. The three-year incidence of fracture in chronic kidney disease. Kidney Int. 2014 Oct;86(4):810-8. doi: 10.1038/ki.2013.547. Epub 2014 Jan 15. PMID 24429401
- [Background] Runesson B, Trevisan M, Iseri K, Qureshi AR, Lindholm B, Barany P, Elinder CG, Carrero JJ. Fractures and their sequelae in non-dialysis-dependent chronic kidney disease: the Stockholm CREAtinine Measurement project. Nephrol Dial Transplant. 2020 Nov 1;35(11):1908-1915. doi: 10.1093/ndt/gfz142. PMID 31361316
- [Background] Kim SM, Long J, Montez-Rath M, Leonard M, Chertow GM. Hip Fracture in Patients With Non-Dialysis-Requiring Chronic Kidney Disease. J Bone Miner Res. 2016 Oct;31(10):1803-1809. doi: 10.1002/jbmr.2862. Epub 2016 Jul 11. PMID 27145189
- [Background] Vilaca T, Salam S, Schini M, Harnan S, Sutton A, Poku E, Allen IE, Cummings SR, Eastell R. Risks of Hip and Nonvertebral Fractures in Patients With CKD G3a-G5D: A Systematic Review and Meta-analysis. Am J Kidney Dis. 2020 Oct;76(4):521-532. doi: 10.1053/j.ajkd.2020.02.450. Epub 2020 Jul 9. PMID 32654892
- [Background] Isakova T, Cai X, Lee J, Mehta R, Zhang X, Yang W, Nessel L, Anderson AH, Lo J, Porter A, Nunes JW, Negrea L, Hamm L, Horwitz E, Chen J, Scialla JJ, de Boer IH, Leonard MB, Feldman HI, Wolf M; CRIC Study Investigators. Longitudinal Evolution of Markers of Mineral Metabolism in Patients With CKD: The Chronic Renal Insufficiency Cohort (CRIC) Study. Am J Kidney Dis. 2020 Feb;75(2):235-244. doi: 10.1053/j.ajkd.2019.07.022. Epub 2019 Oct 23. PMID 31668375
- [Background] Burlacu A, Genovesi S, Goldsmith D, Rossignol P, Ortiz A, Kalra PA, Malyszko J, Banach M, Kanbay M, Covic A. Bleeding in advanced CKD patients on antithrombotic medication - A critical appraisal. Pharmacol Res. 2018 Mar;129:535-543. doi: 10.1016/j.phrs.2017.12.004. Epub 2017 Dec 5. PMID 29208494
- [Background] Flevas DA, Megaloikonomos PD, Dimopoulos L, Mitsiokapa E, Koulouvaris P, Mavrogenis AF. Thromboembolism prophylaxis in orthopaedics: an update. EFORT Open Rev. 2018 Apr 27;3(4):136-148. doi: 10.1302/2058-5241.3.170018. eCollection 2018 Apr. PMID 29780621
- [Background] Reiss AB, Voloshyna I, De Leon J, Miyawaki N, Mattana J. Cholesterol Metabolism in CKD. Am J Kidney Dis. 2015 Dec;66(6):1071-82. doi: 10.1053/j.ajkd.2015.06.028. Epub 2015 Sep 1. PMID 26337134
- [Background] Morris GK, Henry AP, Preston BJ. Prevention of deep-vein thrombosis by low-dose heparin in patients undergoing total hip replacement. Lancet. 1974 Oct 5;2(7884):797-800. doi: 10.1016/s0140-6736(74)91069-1. No abstract available. PMID 4138248
- [Background] Pellegrini VD Jr, Clement D, Lush-Ehmann C, Keller GS, Evarts CM. The John Charnley Award. Natural history of thromboembolic disease after total hip arthroplasty. Clin Orthop Relat Res. 1996 Dec;(333):27-40. PMID 8981880
- [Background] White RH, Zhou H, Romano PS. Incidence of symptomatic venous thromboembolism after different elective or urgent surgical procedures. Thromb Haemost. 2003 Sep;90(3):446-55. doi: 10.1160/TH03-03-0152. PMID 12958614
- [Background] Santana DC, Emara AK, Orr MN, Klika AK, Higuera CA, Krebs VE, Molloy RM, Piuzzi NS. An Update on Venous Thromboembolism Rates and Prophylaxis in Hip and Knee Arthroplasty in 2020. Medicina (Kaunas). 2020 Aug 19;56(9):416. doi: 10.3390/medicina56090416. PMID 32824931
- [Background] Gould MK, Garcia DA, Wren SM, Karanicolas PJ, Arcelus JI, Heit JA, Samama CM. Prevention of VTE in nonorthopedic surgical patients: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e227S-e277S. doi: 10.1378/chest.11-2297. PMID 22315263
- [Background] Douketis JD, Spyropoulos AC, Murad MH, Arcelus JI, Dager WE, Dunn AS, Fargo RA, Levy JH, Samama CM, Shah SH, Sherwood MW, Tafur AJ, Tang LV, Moores LK. Perioperative Management of Antithrombotic Therapy: An American College of Chest Physicians Clinical Practice Guideline. Chest. 2022 Nov;162(5):e207-e243. doi: 10.1016/j.chest.2022.07.025. Epub 2022 Aug 11. PMID 35964704
- [Background] Krauss ES, Segal A, Dengler N, Cronin M, Pettigrew J, Simonson BG. Utilization of the Caprini Score for Risk Stratification of the Arthroplasty Patient in the Prevention of Postoperative Venous Thrombosis. Semin Thromb Hemost. 2022 Jun;48(4):407-412. doi: 10.1055/s-0042-1742739. Epub 2022 Feb 28. PMID 35226947